CLINICAL TRIAL: NCT04443751
Title: A Phase I, Multicenter, Open-label Study of SHR-1702 in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: A Safety and Efficacy Study of SHR-1702 Monotherapy in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1702-I-102
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: AML; MDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1702 monotherapy (Experimental): SHR-1702 monotherapy, given intravenously (IV); dose escalation and dose expansion.
  Interventions: Drug: SHR-1702

INTERVENTIONS:
Drug: SHR-1702 — SHR-1702 monotherapy, administered IV

SUMMARY:
This study will assess the safety and preliminary efficacy of escalating doses of SHR-1702 monotherapy in relapsed/refractory AML and intermediate-high risk MDS

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. ≥18 years of age.
3. Refractory/Relapsed AML, or failed to achieve complete remission after 2 cycles of induction therapy.
4. Intermediate, High and very high risk MDS according to the revised International Prognostic Scoring System (IPSS-R) who have failed prior therapies, such as azacitidine and decitabine (Scoring≥3.5).
5. Life expectancy≥12 months.
6. With Adequate hematologic and organ function
7. Signed inform consent form

Exclusion Criteria:

1. With a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
2. With significant cardiovascular disease.
3. With a history of autoimmune disease.
4. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
5. Positive test result for human immunodeficiency virus (HIV); Active hepatitis B or hepatitis C.
6. Active or untreated central nervous system (CNS) metastases.
7. Active infection within 2 weeks.
8. Know to be allergic to the ingredients of SHR-1702 injection.
9. Prior allogeneic bone marrow transplantation or solid organ transplant
10. With a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of SHR-1702 monotherapy in patients with AML or MDS. | 6 months

SECONDARY OUTCOMES:
Number of participants with the type, frequency, and severity of adverse events (AEs) as a measure of safety and tolerability of SHR-1702 monotherapy in AML and MDS patients | 2 years
Maximum Concentration (Cmax) of SHR-1702 monotherapy in patients with AML or MDS | 2 years
Minimum Concentration (Cmax) of SHR-1702 monotherapy in patients with AML or MDS | 2 years
Immunogenicity as assessed by the presence of anti-drug antibodies | 2 years
  Anti SHR-1702 antibodies will be tested frequently
Pharmacodynamic profile as assessed by receptor occupancy | 2 years
  SHR-1702 receptor occupation
Objective response rate（ORR）for SHR-1702 in AML based on IWG2003 or high risk MDS based on IWG2006 | 2 years
Best of Response（BOR）for SHR-1702 in AML or high risk MDS | 2 years
Progression-Free Survival（PFS) for SHR-1702 in AML or high risk MDS | 2 years
Overall Survival（OS) for SHR-1702 in AML or high risk MDS | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Blood disease hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No